CLINICAL TRIAL: NCT04754269
Title: Randomized Controlled Trial of an M-health Intervention to Reduce Sweet Beverage Consumption Among Low-income Latino Children
Brief Title: A Mobile Health Intervention to Reduce Sweet Beverage Consumption in Latino Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-30664
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Child Obesity; Child Development
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beverage Intervention (Experimental): Parents will watch a video that promotes optimal beverage practices for young children. Parents will receive that reinforce and expand on the messages in the video.
  Interventions: Behavioral: Beverage Intervention
- Reading Intervention (Experimental): Parents will watch a video that promotes reading to children. Parents will receive text messages that reinforce and expand on the messages in the video.
  Interventions: Behavioral: Reading Intervention

INTERVENTIONS:
Behavioral: Beverage Intervention — Parents will watch a video that promotes optimal beverage practices for young children including discouraging consumption of sugar-sweetened beverages and fruit juice and encouraging consumption of water and unsweetened milk. Parents will receive 24 text messages over a 12 week period that reinforce and expand on the messages in the video.
  Arms: Beverage Intervention
Behavioral: Reading Intervention — Parents will watch a video that promotes reading to children and includes specific ideas and techniques for how to make reading interactive and engaging. Parents will receive 24 text messages over a 12 week period that reinforce and expand on the messages in the video.
  Arms: Reading Intervention

SUMMARY:
Sugar-sweetened beverage consumption is a major contributor to childhood obesity, caries, fatty liver disease, and Type 2 diabetes. Latino children are more likely to consume sugar-sweetened beverages (SSBs) and to suffer from all of the aforementioned conditions. Reading out loud to children from birth through age 5 is critical for the promotion of language and early literacy skills. Children whose parents read aloud to them are more likely to start school with the skills required for early reading success. This is important as reading proficiency in third grade is the best predictor of high school graduation and career success. Latino children are less likely to be read to than non-Hispanic white children and at higher risk of entering kindergarten without critical early literacy skills. Thus, there is a pressing need for interventions to reduce SSB consumption among Latino children as well as interventions that promote reading out loud. Primary care is an optimal setting for such interventions. However, multiple demands on providers' time make it difficult to rely on in-person interventions. For this reason, it is critical to test intervention designs that do not rely directly on health care providers and that can be delivered remotely if needed. The investigators have developed two m-health interventions for Latino parents, one that promotes optimal beverage consumption patterns and one that promotes reading out loud to children. The purpose of this study is to test the impact of these interventions on child beverage intake patterns and the frequency with which parents read to children.

ELIGIBILITY:
Inclusion Criteria:

* Parent identifies child as Latino/a/x
* Child age 1 to 5 (12 to 59 months)
* Parent has a cell phone that can receive text messages
* Parent speak English or Spanish

Exclusion Criteria:

• Child does not feed by mouth

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in 7-day child consumption of sugar-sweetened beverages and 100% fruit juice | Change from baseline to 3-month follow-up
  Parents will report child consumption of sugar-sweetened beverages and 100% fruit juice over previous 7 days in fluid ounces via a verbal questionnaire. The outcome measure will be the summed 7-day total of sugar-sweetened beverages and 100% fruit juice in fluid ounces

SECONDARY OUTCOMES:
Change in 7 day total parent intake of sugar-sweetened beverages | Change from baseline to 3-month follow-up
  Parents will report their own consumption of sugar-sweetened beverages in the previous 7 days in 8 ounce servings via a verbal questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Beck, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital Children's Health Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No